CLINICAL TRIAL: NCT02431104
Title: Clinical Evaluation of Tattoo Removal Using a Novel Dual-Wavelength, Dual-Pulse Duration Laser"
Brief Title: Clinical Evaluation of Tattoo Removal Using a Novel Dual-Wavelength, Dual-Pulse Duration Laser
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study.
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-15-EN02
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Laser Tattoo Removal

ARMS (1):
- Laser Treatment (Experimental): Treatment to unwanted tattoo using a 532-nm KTP/1064-nm Nd:YAG Dual-Pulse Duration Laser
  Interventions: Device: 532-nm KTP/1064-nm Nd:YAG Dual-Pulse Duration Laser

INTERVENTIONS:
Device: 532-nm KTP/1064-nm Nd:YAG Dual-Pulse Duration Laser — Cutera enlighten dual wavelength 532nm KTP/1064nm Nd:YAG laser
  Other Names: Enlighten laser

SUMMARY:
A single-center prospective, open-label, uncontrolled study in 10 male or female subjects, age 18 to 65 years, who desire laser removal of a tattoo which contains all black ink.

DETAILED DESCRIPTION:
This is a single-center prospective, open-label, uncontrolled study in 10 male or female subjects, age 18 to 65 years, who desire laser removal of a tattoo which contains all black ink. Subjects will receive up to 5 laser treatments, spaced 4 to 6 weeks apart, and will be followed at 3 months post-final treatment. Number of laser treatments required shall be based upon tattoo response to laser irradiation. The Investigator will terminate laser treatments upon 100% clearance of tattoo or after 5 treatment sessions, or in the event of an adverse effect which requires cessation of laser treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - VI
* Target tattoo contains only black ink, is more than 1 year old and must have been obtained from a professional tattoo parlor.
* Wiling to cover tattoos with a bandage or clothing; and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated area starting 2 to 4 weeks before the treatment and/or every day for the duration of the study, including the follow-up period.

Exclusion Criteria:

* Target tattoo is 'home made' OR was obtained from an amateur artist.
* Presence of double tattoo in the treatment area or presence of tribal, scarred, high-ink density, or highly colorful single tattoo.
* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* History of allergic reaction to pigments following tattooing.
* History of allergy to local anesthetics.
* History of malignant tumors in the target area.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment of improvement post-final treatment | 3 months
  Assessment of tattoo clearance by independent blinded reviewers

SECONDARY OUTCOMES:
Subject's Global Assessment of improvement post-final treatment | 3 months
  Assessment of tattoo clearance by subject
Subject Satisfaction post-final treatment | 3 months
  Assessment of subject satisfaction with treatment results.
Incidence and severity of adverse device effects | Day 0, 4 wks, 8wks, 12 wks, 16 wks, 28 wks
  Assessment of ADEs immediately following each laser treatment and at the final follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Sapra, MD, Principal Investigator — ICLS Dermatology and Plastic Surgery
Locations (1):
- ICLS Dermatology and Plastic Surgery, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No